CLINICAL TRIAL: NCT03539991
Title: SWOG Tobacco Program for the Oncology Practice
Brief Title: Developing an eLearning Program in Helping Spanish and Portuguese Speaking Cancer Care Providers During Tobacco Use Counselling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PA17-0878; NCI-2018-01340 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA17-0878 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-05-16; First posted 2018-05-30 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Health Care Provider

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (online course, virtual meeting) (Experimental): Participants complete an online course focusing on different aspects of tobacco prevention and cessation over 1 hour each per week for 4 weeks. They also engage in 6 virtual meetings over 1 hour about tobacco use once per month.
  Interventions: Other: Internet-Based Intervention; Other: Meeting; Other: Survey Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Complete online courses
Other: Meeting — Participate in virtual meetings
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial aims to develop an electronic learning (eLearning) program and mobile tool for Spanish and Portuguese speaking cancer care providers to use in tobacco counseling of their patients. This study may provide information for the design and implementation of tobacco cessation training programs directed to this group of professionals in low- and middle-income countries for the Latin American region.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop and test the feasibility of an eLearning program on brief tobacco counseling specifically designed for Spanish- and Portuguese-speaking cancer care providers.

II. To linguistically/culturally tailor and test a mobile tool designed to assist in providing effective tobacco counseling and treatment.

OUTLINE:

Participants complete an online course focusing on different aspects of tobacco prevention and cessation over 1 hour each per week for 4 weeks. They also engage in 6 virtual meetings over 1 hour about tobacco use once per month.

After completion of study, participants are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Be a cancer care provider (CCP) working at one of the above cancer centers
* Have direct contact with cancer patients
* Have access to the internet during the 4-hour online course and at least once per month to participate in post-training virtual meetings, discussion board postings, email, and periodic audio chat conferences
* Have access to a computer, tablet, or smartphone (iPhone or Android) with built-in camera and microphone
* Have basic proficiency in the use of a computer, including word processing and email
* Commit to the STOP Program by completing the online course and sharing lessons learned with other CCPs at the monthly virtual meetings that will take place during the 6 months following course completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention rates | Up to 6 months
  Will be used as key parameters for assessing the feasibility of the eLearning program. The Wilcoxon signed-rank test will be used to compare scores obtained in the pre- and post-tests of the eLearning program. Effect sizes will be computed as the absolute value of the difference between the post-test (T2, T3, and T4) and pre-test (T1) scores divided by the mean of the standard deviations for each.
Linguistically/culturally tailored mobile tool | Up to 6 months
  Computing the System Usability Scale (SUS) scores in the final assessment will allow our research team to analyze cancer care provider's (CCPs) experience of using the tool. A descriptive analysis to compute the SUS score will be performed and later converted to percentile ranks. A percentile rank of 75% will indicate that the tool has high perceived usability. All statistical analyses will be performed using SPSS Statistics version 23 (International Business Machines Corporation).

OTHER OUTCOMES:
Gains in participants' competencies in providing smoking cessation assistance to cancer patients | Baseline up to 6 months
  Will be assessed by comparing pre- and post-test responses to the International Association for the Study of Lung Cancer survey. Item distributions, mean, median, standard deviation, minimum, maximum, and skewness will be explored. Skewness values between -1 and 1 will be considered acceptable. To examine reliability and internal consistency of each of the items assessing cancer care providers CCPs' competency for providing brief tobacco counseling, Cronbach's alphas will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- Hosptial de Cancer de Barretos, Barretos, São Paulo, Brazil
- Instituto Nacional De Cancerologia, Bogotá, Colombia
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org